CLINICAL TRIAL: NCT07188909
Title: Clinical Observation on the Efficacy of Patient-Donor Derived Probiotics in Improving Intestinal Flora Disorder in Patients With Intestinal Acute Graft-Versus-Host Disease (aGVHD)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025086
Record Dates: First submitted 2025-08-26; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Acute Graft-Versus-Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient-Donor Derived Probiotics (Experimental): To clinically evaluate the efficacy of patient- and/or donor-derived probiotics in ameliorating intestinal flora dysbiosis in patients with acute intestinal graft-versus-host disease (aGVHD), thereby mechanistically enhancing clinical outcomes and quality of life through intestinal microbiome modulation.
  Interventions: Drug: Patient-Donor Derived Probiotics

INTERVENTIONS:
Drug: Patient-Donor Derived Probiotics — To clinically evaluate the efficacy of patient- and/or donor-derived probiotics in ameliorating intestinal flora dysbiosis in patients with acute intestinal graft-versus-host disease (aGVHD), thereby mechanistically enhancing clinical outcomes and quality of life through intestinal microbiome modulation.

SUMMARY:
To clinically evaluate the efficacy of patient- and/or donor-derived probiotics in ameliorating intestinal flora dysbiosis in patients with acute intestinal graft-versus-host disease (aGVHD), thereby mechanistically enhancing clinical outcomes and quality of life through intestinal microbiome modulation.

DETAILED DESCRIPTION:
Study Design Overview:

Ten patients aged >50 years scheduled for haploidentical hematopoietic stem cell transplantation (HSCT) will be enrolled. Stool specimens will be collected from both patients and donors (due to frequent depletion of beneficial bacteria in such patients, donor specimens are essential to enhance probiotic detection and cultivation rates). Patient specimens will undergo 16S rDNA intestinal microbiome analysis.

Upon clinical diagnosis of intestinal aGVHD:

1. Pre-collected patient and donor specimens will be homogenized
2. Target isolation and culture of core beneficial bacteria (Lactobacillus and Bifidobacterium)
3. Strain identification via TOF mass spectrometry
4. Fermentation and preparation of 200 enteric-coated capsules (100 Lactobacillus capsules + 100 Bifidobacterium capsules)

Post-intervention assessment (100 days after administration):

Changes in microbiome composition, relative abundance, species diversity, biochemical indicators, and bowel movement characteristics will be evaluated to assess the therapeutic efficacy of patient/donor-derived Lactobacillus and Bifidobacterium in GVHD.

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible for this study must satisfy all of the following criteria:

1. Age >50 years, regardless of gender;
2. Scheduled for haploidentical hematopoietic stem cell transplantation;
3. ECOG performance status score ≤2;
4. Voluntarily participate and provide written informed consent.

Exclusion Criteria:

Subjects presenting with any of the following conditions will be excluded from this study:

1. Active or chronic infectious diseases, including recent febrile symptoms (axillary temperature ≥37.3°C within 48h);
2. Gastrointestinal disorders:

   * Clostridioides difficile infection (CDI): Recurrent or refractory CDI;
   * Other conditions: Ulcerative colitis, Crohn's disease, irritable bowel syndrome (IBS), diarrhea associated with dysbiosis, liver cirrhosis;
3. Allergic or immune-mediated diseases:

   Autoimmune hepatitis, systemic lupus erythematosus (SLE), ankylosing spondylitis, immune-mediated osteoarthritis, allergic dermatitis, immune thrombocytopenic purpura (ITP);
4. Antibiotic usage within 7 days prior to enrollment.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-03-04 (Estimated); Study Completion 2026-03-04 (Estimated)

PRIMARY OUTCOMES:
Clinical response rate of intestinal acute graft-versus-host disease (aGVHD) | within 100 days
  Changes of stool frequency of subjects before and after taking probiotic capsules from patients.

SECONDARY OUTCOMES:
To study the changes of intestinal flora of subjects before and after taking probiotics from patients for 100 days | within 100 days
  16SrDNA intestinal flora detection, to study the changes of Bifidobacterium, Lactobacillus and Clostridium before and after taking probiotics from patients for 100 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Tianjin, Tianjin Municipality, China